CLINICAL TRIAL: NCT02723162
Title: Translational Neuropsychopharmacology Research of Nicotine Addiction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Gray, MD, Pricipal Investigator - Medical, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: PRO#48152
Record Dates: First submitted 2016-03-07; First posted 2016-03-30 (Estimated); Results first posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: Nicotine Dependence, Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VRN+ NAC (Experimental): Titrated VRN up to 1mg BID with NAC at 1200mg BID for 28 days
  Interventions: Drug: Varenicline (VRN); Drug: N-Acetylcysteine (NAC)
- NAC+ PBO (Active Comparator): 1200mg BID for 28 days plus VRN placebo for 28 days
  Interventions: Drug: N-Acetylcysteine (NAC); Drug: Placebo
- VRN+ PBO (Active Comparator): Titrated VRN up to 1mg BID with NAC placebo for 28 days
  Interventions: Drug: Varenicline (VRN); Drug: Placebo
- PBO+PBO (Placebo Comparator): Double placebo taken for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline (VRN) — VRN will be provided at the standard recommended dose (0.5 mg daily for 3 days, then 0.5 mg twice daily for 4 days, then 1 mg twice daily thereafter for the remaining 21 days of active treatment.
  Arms: VRN+ NAC; VRN+ PBO
Drug: N-Acetylcysteine (NAC) — NAC will be dosed at 1200 mg twice daily throughout the 28-day active treatment
  Arms: NAC+ PBO; VRN+ NAC
Drug: Placebo — Matched placebo
  Arms: NAC+ PBO; PBO+PBO; VRN+ PBO

SUMMARY:
This study will examine the effects of combining Varenicline (VRN) and N-acetylcysteine (NAC) on neural circuitry function and treating nicotine addiction. Healthy adult nicotine dependent cigarette smokers interested in quitting (n=110) will be randomized to one of four PBO-controlled conditions for 4 weeks: 1) VRN+NAC, 2) VRN+PBO, 3) NAC+PBO or 4) PBO+PBO. Following 1 week of medication, participants will be contingently reinforced for 3 days of smoking abstinence and be scanned using functional magnetic resonance imaging (fMRI) techniques, while nicotine deprived during a resting state and a cue-reactivity (CR) task. Participants will be followed over the next 3 weeks of treatment and clinical variables will be assessed.

DETAILED DESCRIPTION:
Cigarette (henceforth nicotine) addiction is a chronic, relapsing brain disorder and remains the leading preventable cause of death and disability in the US, costing nearly $200 billion each year. Although ~20% of adults in the USA currently smoke, the majority want to quit. In spite of the breadth of research focused on improving health outcomes and reducing the societal burden caused by nicotine addiction, the majority of smokers who attempt to quit will relapse. Nicotine withdrawal-related disturbances in executive function, negative affect and reward processes compel a smoker to self-administer nicotine-each in turn representing the loss of control to remain abstinent and risk factors for relapse. Thus, identifying the effects of nicotine addiction on mechanisms of self-regulation, and the value of novel medications for remediating dysregulated behavior are both needed in order to enhance interventions for treating nicotine addiction. The preliminary data, along with the extant literature, suggest that the maintenance of nicotine addiction is subserved by dysregulated neural function in limbic-striatal and corticostriatal neural circuitry. While VRN may be effective in treating limbic-striatal circuitry that is associated with promoting abstinence and reducing acute withdrawal; NAC may be effective in treating corticostriatal circuitry function that is associated with relapse vulnerability. Thus, the current proposal seeks to investigate two medications (VRN & NAC), with potentially complementary effects on the two different brain circuits- limbic-striatal (VRN) and corticostriatal (NAC) circuitry-and that may therapeutically target two different phases in the recovery of nicotine addiction-the promotion of abstinence (VRN) and relapse prevention (NAC). The placebo (PBO)-controlled design in this proposal will allow the team to identify and translate between the neurobiological substrates and the neurocognitive underpinnings of the effects of VRN+NAC on smoking behavior in humans-thus, advancing the understanding of the pathophysiology of nicotine addiction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 55
2. Right Handed
3. English fluency
4. 20/20 vision with corrective lenses.
5. Smoke ≥ 10 cigarettes/day for a minimum of two years and have an expired carbon monoxide (CO) concentration of ≥ 10 ppm (to confirm inhalation).
6. Interest in quitting smoking or contemplating a quit attempt in the next 6 months
7. If female, agreement to use birth control

Exclusion Criteria:

1. Past head injury or primary neurological disorder associated with MRI abnormalities, including dementia, MCI, brain tumors, epilepsy, Parkinson's disease, or demyelinating diseases
2. Any physical or intellectual disability affecting completion of assessments
3. Any contraindication to MRI
4. Positive urine drug screen for illicit substances (such as marijuana or cocaine).
5. Current or past psychosis
6. Electroconvulsive therapy in last 6 months
7. Use of antidepressant medications or other psychotropic medications in the last month.
8. Positive urine pregnancy test or current breast feeding status

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VRN+ NAC | NAC+ PBO | VRN+ PBO | PBO+PBO
Started | 18 | 15 | 17 | 17
Day 10 fMRI Visit | 15 | 11 | 14 | 15
Completed | 12 | 10 | 13 | 12
Not Completed | 6 | 5 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRN+ NAC | NAC+ PBO | VRN+ PBO | PBO+PBO | Total
Number analyzed (Participants) | 18 | 15 | 17 | 17 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 17 | 17 | 67
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (8.9) | 35.1 (12.8) | 42.4 (9.8) | 37.1 (9.6) | 39.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 8 | 31
  Male | 10 | 8 | 9 | 9 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 18 | 13 | 16 | 16 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 3 | 3 | 20
  White | 12 | 7 | 12 | 13 | 44
  More than one race | 0 | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 17 | 17 | 67
Cigarettes Smoked Per Day [Mean (Standard Deviation); unit: Cigarettes Per Day] | 16.8 (12.6) | 13.7 (10.4) | 17.3 (11.4) | 20.0 (19.2) | 17.3 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Blood Oxygen Level Dependent (BOLD) Signal Response
Description: Measure the Effects of Varenicline and N-Acetylcysteine (NAC) on brain activation to smoking images while participants undergo Functional Magnetic Resonance (fMRI) Imaging. Mean percent signal change of fMRI BOLD in the insula and nucleus accumbens will be recorded during smoking images. The lower the BOLD signal response, the better the outcome, meaning reduced reactivity to smoking images.
Time Frame: 10 Days
Measure: Median (Inter-Quartile Range); unit: Percentage change
Arm/Group | VRN+ NAC | NAC+ PBO | VRN+ PBO | PBO+PBO
Number analyzed (Participants) | 15 | 11 | 14 | 15
Percentage change
  Insula | -0.09 [-1.14 to 0.77] | 1.07 [0.39 to 1.41] | 0.08 [-0.36 to 0.33] | 1.19 [0.78 to 2.84]
  Nucleus Accumbens | 0.11 [-0.25 to 0.67] | 0.91 [-0.15 to 1.81] | 0.12 [-0.81 to 1.10] | 1.43 [0.94 to 2.25]

2. Primary Outcome: rZ Change Score in Resting State Functional Connectivity From Baseline
Description: Measure the effects of Varenicline and N-Acetylcysteine on resting-state functional connectivity while participants undergo fMRI. Fisher transformed correlation (rZ) scores will be recorded between medial prefrontal cortex and ventral striatum during a resting state scan. The higher the rZ score, the better the outcome, meaning stronger functional connectivity. rZ scores range from -1 to 1. The rZ-score central value is analogous to a central value to of a Z-score of 0, representing the population mean.
Time Frame: Baseline to day 10
Measure: Median (Standard Error); unit: Fisher Z
Arm/Group | VRN+ NAC | NAC+ PBO | VRN+ PBO | PBO+PBO
Number analyzed (Participants) | 16 | 14 | 11 | 15
Fisher Z | .297 (.053) | .060 (.042) | .181 (.053) | .191 (.058)

3. Secondary Outcome: Number of Cigarettes Smoked Per Day
Description: Measure the effects of Varenicline and N-Acetylcysteine on smoking behavior over the course of the study
Time Frame: 28 Days
Population: Analysis population consists of randomized participants that had data available at study day 7 or beyond.
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | VRN+ NAC | NAC+ PBO | VRN+ PBO | PBO+PBO
Number analyzed (Participants) | 15 | 13 | 14 | 16
Cigarettes per day | 5.3 (5.5) | 4.0 (4.8) | 5.3 (3.9) | 5.0 (4.5)

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | VRN+ NAC | NAC+ PBO | VRN+ PBO | PBO+PBO
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/17 | 2/17
Other Adverse Events (participants affected / at risk) | 4/18 | 5/15 | 3/17 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRN+ NAC (N=18) | NAC+ PBO (N=15) | VRN+ PBO (N=17) | PBO+PBO (N=17)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1)
Choleithiasis (worsening) (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRN+ NAC (N=18) | NAC+ PBO (N=15) | VRN+ PBO (N=17) | PBO+PBO (N=17)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (5)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Eye Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Worsening) (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Increased Energy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post Operative Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash, Generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnambulism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (worsening) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Poor Quality Sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-Traumatic Pain (Worsening) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychological Trauma (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study did not reach full planned enrollment due to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02723162/Prot_SAP_000.pdf